CLINICAL TRIAL: NCT06618274
Title: Navigation and Research: Evaluating the Intervention of Central Navigation and an Oncology Research Navigator (ORN) on Cancer Outcomes and Clinical Trial Enrollment (NAVIGATE Trial)
Brief Title: Effectiveness of Central Oncology Navigation and the Use of an ORN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC2334
Record Dates: First submitted 2024-09-25; First posted 2024-10-01 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Malignant Tumor
Keywords: navigation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Cohort 1 will enroll patients with new cancer appointments within genitourinary (GU) or thoracic cancers. These clinics have not yet implemented the central navigation program.
  Interventions: Behavioral: Central oncology navigation (SOC)
- Cohort 2 (Experimental): Cohort 2 will enroll participants with new cancer appointments within gastrointestinal (GI), hematology, and breast cancer (clinics where the central navigation program was implemented). These individuals will be randomized to receive standard of care, which for these cancer types includes central oncology navigation or the intervention of oncology research navigator in addition to SOC.
  Interventions: Behavioral: Intervention of oncology research navigator embedded in central oncology navigation

INTERVENTIONS:
Behavioral: Intervention of oncology research navigator embedded in central oncology navigation — The intervention of oncology research navigator or Oncology research navigator (ORN) is embedded in central oncology navigation cancer care delivery.
  Other Names: oncology research navigator (ORN
  Arms: Cohort 2
Behavioral: Central oncology navigation (SOC) — Central oncology navigation (SOC ) alone.
  Arms: Cohort 1

SUMMARY:
This health services interventional study investigates the effectiveness of central oncology navigation (SOC ) alone and central oncology navigation with a new role called an "oncology research navigator (ORN)" who is embedded in central oncology navigation cancer care delivery. This study will examine two patient cohorts: Cohort 1 will enroll patients with new cancer appointments within genitourinary (GU) or thoracic cancers. These clinics have not yet implemented the central navigation program. Participants will be enrolled pre- and post-implementation of the central oncology navigator within these cancer groups to evaluate the effectiveness of the central oncology navigator alone. The second cohort will enroll participants with new cancer appointments within gastrointestinal (GI), hematology, and breast cancer (clinics where the central navigation program was implemented). These individuals will be randomized to receive standard of care, which for these cancer types includes central oncology navigation or the intervention of an oncology research navigator in addition to SOC. This intervention will involve baseline and biweekly follow-up for a total of 3 months. Interactions with the ORN will include facilitating participation in supportive care services and clinical trials. All participants will undergo baseline and follow-up patient-reported outcomes and data collection. The study will evaluate the impact of the central oncology navigation program alone, as well as the addition of the ORN on patient quality of life, as well as enrollment into studies and participation in supportive care services. Additional analyses will evaluate the impact of the central oncology navigation program on patient experience, patient activation, net promoter scores, and overall survival.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in this study a subject must meet all of the eligibility criteria outlined below.

* Informed consent obtained to participate in the study and HIPAA authorization for release of personal health information.
* Subject is willing and able to comply with study activities based on the judgement of the investigator.
* Age ≥ 18 years at the time of consent.
* Subject has a new patient appointment for cancer care at a UNC Medical Center and a confirmed cancer diagnosis.

Exclusion Criteria:

* Lack of internet access.
* Inability to understand the English language.
* Psychological or other disability resulting in the inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 686 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2027-01-10 (Estimated); Study Completion 2031-07-01 (Estimated)

PRIMARY OUTCOMES:
Cohort 1-supportive service offered | Up to 6 months
  Participation in at least 1 supportive service offered will be measured by the number of patients receiving services. This information will be gathered from chart review.
Cohort 2: number of patients enrolled | Up to 6 months
  Enrollment into non-treatment clinical studies will be measured by the number of patients enrolled at any time. This information will be gathered from chart review.

SECONDARY OUTCOMES:
Cohort 1: Health-related quality of life | Baseline and 3 months
  Cohort 1: Health-related quality of life will be measured using the PROMIS Global Health. The PROMIS Global Health is a comprehensive tool designed to assess an individual's overall physical, mental, and social health and includes 10 items that cover various health domains. These items are divided into two main components: Global Physical Health and Global Mental Health. Global Physical Health: This includes items related to physical functioning, pain, fatigue, and overall physical health. Global Mental Health: This includes items related to mental health, emotional distress, and social health.Response Options: Each item is rated on a 5-point Likert scale, with higher scores indicating better health.Raw Scores: The responses are summed to create raw scores for both the Global Physical Health and Global Mental Health components.
Cohort 1: Patient activation | Baseline and 3 months
  Cohort 1: Patient activation will be measured using Patient Activation Measure -13 (PAM-13). PAM-13 is a validated questionnaire designed to assess an individual's knowledge, skills, and confidence in managing their own health and healthcare. It consists of 13 items that measure patient activation, which is the extent to which individuals feel capable of managing their health. The PAM 13 includes 13 statements that respondents rate based on their level of agreement, ranging from "Strongly Disagree" to "Strongly Agree." Responses are scored on a scale from 0 to 100. Higher scores indicate greater patient activation.
Cohort 1: Patient experience | Baseline and 3 months
  Cohort 1: Patient experience will be measured using the Consumer Assessment of Healthcare Providers and Systems (CAHPs) cancer care survey. Scoring will be any number from 0 to 10, where 0 is the worst cancer care team possible and 10 is the best cancer care team possible, what number would you use to rate your cancer care team? (0-10 rating, from "worst cancer care team possible" to "best cancer care team possible" 2. Considering all your cancer care at this cancer center, using any number from 0 to 10, where 0 is the worst overall cancer care experience possible and 10 is the best overall cancer care experience possible, what number would you use to rate your overall cancer care experience? (0-10 rating, from "worst overall cancer care experience possible" to "best overall cancer care experience possible")
Cohort 1: Net promoter | Baseline and 3 months
  Cohort 1: Net promoter scores will be measured using the net promoter score survey.
  The Net Promoter Score (NPS) is used as a metric for assessing customer loyalty and satisfaction. NPS measures the likelihood of customers to recommend a company's product or service to others. It is based on a single question: "On a scale from 0 to 10, how likely are you to recommend our product/service to a friend or colleague?"
Cohort 1: Overall Survival | Up to 5 years
  Cohort 1: Overall Survival, defined as death by any cause from the time of enrollment will be measured. Any patient who has not died by the analysis date will be censored. Sub-analyses for cancer types will be conducted.
Cohort 2: Health-related quality of life | Baseline and 3 months
  Cohort 2: Health-related quality of life will be measured using the PROMIS Global Health 10-item instrument in all participants The PROMIS Global Health is a comprehensive tool designed to assess an individual's overall physical, mental, and social health and includes 10 items that cover various health domains. These items are divided into two main components: Global Physical Health and Global Mental Health. Global Physical Health: This includes items related to physical functioning, pain, fatigue, and overall physical health. Global Mental Health: This includes items related to mental health, emotional distress, and social health.Response Options: Each item is rated on a 5-point Likert scale, with higher scores indicating better health.Raw Scores: The responses are summed to create raw scores for both the Global Physical Health and Global Mental Health components.

CONTACTS AND LOCATIONS:
Overall Officials: William A Wood, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials